CLINICAL TRIAL: NCT06766799
Title: Comparison Between Handheld Rebound Tonometer and Applanation Tonometer in IOP Measurement in Paediatric Glaucomas
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Norhan Alateek Foaad, Resident Doctor, Sohag University
Other Study IDs: Soh-Med-2025
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A ( Glaucomatous Patients)
  Interventions: Device: Rebound and Applanation Tonometer
- Group B ( Control Group)
  Interventions: Device: Rebound and Applanation Tonometer

INTERVENTIONS:
Device: Rebound and Applanation Tonometer — Measurement of Intraocular Pressure

SUMMARY:
To compare the accuracy between handheld rebound tonometer & applanation tonometer in IOP measurement in pediatric glaucoma cases

ELIGIBILITY:
Inclusion Criteria:

* Patients attending to our pediatric glaucoma clinic diagnosed with glaucoma aged >18 years old are subjected to IOP Measurements.

Exclusion Criteria:

* **Patients aged more than 18 years old

  * patients with scarred cornea

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 100 Cases of Glaucomatous Patients and 60 Cases of Healthy Individuals
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between the IOP Measurments by Rebound Tonometer & Applanation tonometer | over nine months
  To compare the accuracy between handheld rebound tonometer & applanation tonometer in IOP measurement in pediatric glaucoma cases